CLINICAL TRIAL: NCT01698476
Title: Immune Reconstitution in Tuberculosis Disease Using Antimicrobial Treatment With Vitamin D and Phenylbutyrate
Brief Title: Immune Reconstitution in Tuberculosis Disease
Acronym: IRETB
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Addis Ababa University (Other); Armauer Hansen Research Institute, Ethiopia (Other)
Responsible Party: Principal Investigator, Susanna Brighenti, Associate professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRETB-2012
Record Dates: First submitted 2012-09-25; First posted 2012-10-03 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-02

CONDITIONS: Pulmonary Tuberculosis (TB)
Keywords: pulmonary TB; cholecalciferol; sodium phenylbutyrate; antimicrobial peptides; immune response
MeSH Terms: conditions — Tuberculosis, Pulmonary | interventions — Vitamin D; Cholecalciferol; 4-phenylbutyric acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- vitamin D (cholecalciferol) and PBA (sodium phenylbutyrate) (Active Comparator): Dose of interventions: 5,000 IU of vitamin D (cholecalciferol tablets) once daily and 500 mg PBA (sodium phenylbutyrate tablets) twice daily for 16 weeks.
  Interventions: Drug: vitamin D (cholecalciferol) and PBA (sodium phenylbutyrate)
- Placebo tablets (Placebo Comparator): Placebo tablets for vitamin D once daily and placebo tablets for PBA (phenylbutyrate) twice daily for 16 weeks.
  Interventions: Drug: Placebo tablets

INTERVENTIONS:
Drug: vitamin D (cholecalciferol) and PBA (sodium phenylbutyrate) — Dose of interventions: 5,000 IU of vitamin D (cholecalciferol tablets) once daily and 500 mg PBA (sodium phenylbutyrate tablets) twice daily for 16 weeks.
  Arms: vitamin D (cholecalciferol) and PBA (sodium phenylbutyrate)
Drug: Placebo tablets
  Arms: Placebo tablets

SUMMARY:
The aim with study is to provide adjunctive therapy with vitamin D and phenylbutyrate together with standard anti-tuberculosis treatment to significantly improve clinical recovery among patients with untreated, active pulmonary tuberculosis.

ELIGIBILITY:
Inclusion Criteria:

HIV negative patients, adult patients >18 years who has not started anti-TB therapy.

Newly diagnosed pulmonary TB confirmed by microscopy or culture but also sputum-negative clinical TB cases (defined according to the WHO 2006 criteria for sputum smear-negative TB ie. clinical symptoms of TB, chest X-ray findings and response to standard treatment).

Exclusion Criteria:

Patients who have already started treatment with anti-TB drugs for more that 5 days.

HIV-positive patients.

History of anti-TB treatment in the past 2 years.

Local extra-pulmonary TB in the absence of lung manifestations.

Hypercalcaemia (serum calcium > 3 mmol/L) identified at baseline.

Pregnant and breast feeding women.

Any known liver or kidney function abnormality, malignancy or patients treated with cardiac glycosides.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Actual)
Dates: Start 2012-09; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Composite clinical TB score | 0 (baseline) compared to 8 weeks.
  A previously described composite clinical TB score will be used to monitor the efficacy of vitamin D and phenylbutyrate treatment among TB patients on standard chemotherapy. The numerical TB score will include self-reported clinical symptoms (cough, night sweats and chest pain) as well as different parameters determined upon clinical examination anemia, haemoptysis, dyspnoea, tachycardia, positive finding at lung auscultation, fever, low body mass index (BMI) and low mid upper arm circumference (MUAC). The TB score will be determined at the time of diagnosis (time point 0) and at 4, 8, 16 and 24 weeks after initiation of antimicrobial treatment with vitamin D and phenylbutyrate. The primary endpoint will be assessed at time point 8 weeks compared to baseline (time point 0).

SECONDARY OUTCOMES:
Clinical secondary endpoints | 0-4, 8, 16 and 24 weeks
  Clinical composite TB score (0, 4, 16, 24 weeks).
  Modified clinical composite TB score (0, 4, 8, 16, 24 weeks).
  Chest X-ray (0, 4, 8, 16, 24 weeks).
  Time to sputum- and/or TB culture conversion (0, 1, 2, 3, 4, 8 weeks).
Laboratory secondary endpoints | 0, 4, 8, 16, 24 weeks
  Peripheral CD4/CD8 T cell counts.
  Antibodies in lymphocytes secertions (ALS) (S Ashenafi, Thorax, 2012).
  Quantiferon-in-tube TB-gold (QFT).
  Plasma levels of vitamin D, LL-37 and also cytokine/chemokine profiles.
  Functional studies of immune cells (PBMCs).

CONTACTS AND LOCATIONS:
Overall Officials: Susanna Brighenti, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Black Lion Hospital (BLH), Addis Ababa University, Faculty of Medicine, Addis Ababa, Lideta Sub City, Ethiopia

REFERENCES:
- [Derived] Bekele A, Gebreselassie N, Ashenafi S, Kassa E, Aseffa G, Amogne W, Getachew M, Aseffa A, Worku A, Raqib R, Agerberth B, Hammar U, Bergman P, Aderaye G, Andersson J, Brighenti S. Daily adjunctive therapy with vitamin D3 and phenylbutyrate supports clinical recovery from pulmonary tuberculosis: a randomized controlled trial in Ethiopia. J Intern Med. 2018 Sep;284(3):292-306. doi: 10.1111/joim.12767. Epub 2018 May 23. PMID 29696707